CLINICAL TRIAL: NCT02481895
Title: Efficacy of an Innovative E-neurocognitive Module as Adjunct to Functional Remediation for Bipolar Disorder
Brief Title: Efficacy of an Innovative E-neurocognitive Module for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22039
Record Dates: First submitted 2015-06-24; First posted 2015-06-25 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder
Keywords: cognition; psychosocial functioning
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): E-neurocognitive module training.
  Interventions: Behavioral: E-neurocognitive module
- Control (No Intervention): The group will note receive any sort of add-on training, just the recommendations from the therapists.

INTERVENTIONS:
Behavioral: E-neurocognitive module — The experimental group will take part of a 12-week extension with a total of 36 hours training with the e-neurocognitive module tailored for bipolar patients
  Arms: Experimental

SUMMARY:
Between 40% and 60% bipolar patients experience neurocognitive impairment not only during acute mood episodes but also during remission periods. These rates are quite similar to those reported as regards to functional impairment. In fact, it is estimated that only one third of patients achieve full social and occupational recovery and get back to their premorbid levels. Moreover, neurocognitive deficits, together with other clinical and sociodemographic variables are thought to contribute to functional impairment for bipolar disorder, similarly to that found in schizophrenia. Little is published with regard to neurocognitive remediation in bipolar disorder. The first open label study on bipolar disorder was published in 2010 with positive results. Recently, a multicenter randomized clinical trial coordinated showed efficacy of an innovative intervention at improving functioning and reducing disability of bipolar patients. There is a need of investigating novel and creative ways to work on cognitive deficits including new technologies in order to reduce costs and increasing benefits for patients. No study addressing computerized cognitive training in bipolar disorder has been developed so far. This project aims to test the efficacy of an e-neurocognitive module as an adjunct to functional remediation in bipolar patients.

DETAILED DESCRIPTION:
This is a randomized clinical study, rater-blind, placebo-controlled stratified by age, sex and educational level to assess the efficacy of a new program, an adjunctive e-neurocognitive module, to functional remediation intervention. The primary outcome measure will be the improvement in global psychosocial functioning measured blindly as the mean change in score Functioning Assessment Short Test from baseline to endpoint. The sample will be composed by 132 euthymic bipolar (type I or II) patients who will be assessed at baseline regarding several clinical, functional and neuropsychological variables. Subsequently, the patients will consecutively start the functional remediation groups, once the group will be finished the patients will be randomly assigned (1:1) to two different groups. The experimental group (EG, 66 patients) will take part of a 12-week extension with a total of 36 hours training with the e-cognitive module tailored for bipolar patients whilst the control group (CG, 66 patients) will not receive any sort of add-on training just the recommendations from the therapists to train the same amount of time that the experimental group: twice per week a total of 3 hours with the material provided during the functional remediation group. All patients will keep on receiving standard psychiatric treatment according to the local treatment guidelines for the management of bipolar patients. At nine months, once the home training has been completed, all patients will be assessed again regarding several clinical, functional and neuropsychological variables. All patients will be assessed monthly regarding several clinical variables, including mood measurements (YMRS and HDRS). At 24 months from baseline, all measurements will be repeated to all patients. In total, three assessments will be conducted (baseline, post-intervention and at 2 years follow-up). The first active intervention that all patients will be receiving is the Functional Remediation Program:

* The Functional Remediation Program which consists of 21 weekly sessions, 90 minutes each. This intervention addresses neurocognitive issues such as attention, memory and executive functions but focuses even more on enhancing functioning in daily routine. The content of this intervention is based on ecological tasks to be performed in two settings, in the clinical but also at home. Patients were trained with exercises in memory, attention, problem solving and reasoning, multitasking and organization in order to improve their functional outcome. Most of the techniques were based on "paper and pencil" tasks and group activities.

After the randomization some patients will continue their training through an e-neurocognitive module specially adaptated for bipolar patients.

1. The e- neurocognitive module will be tailored to bipolar patient's cognitive and functional profile using a newly developed personalized and cost effective technology adapted from a program that has been applied to patients with acquired brain injury. The total duration will be of 36 hours distributed as 1'5 hours twice per week with the aim to enhance cognitive impairment and functioning using a flexible system (website). Therefore, the novelty of this current project is that this is the first trial to test the implementation of an innovative neurocognitive intervention for bipolar patients and its impact on daily life, using new technologies, reducing stigma, transferring responsibilities to the patient, providing the opportunity to improve cognitive deficits at home, being monitored by a neuropsychologist from the hospital, with a good balance costs-benefits. The emphasis will stress on social cognition skills which are highly correlated with psychosocial functioning.
2. Control group. Will receive standard instructions once finished the functional remediation group in order to keep training at home.

In the two groups pharmacological treatment will be prescribed according to the local treatment guidelines for the management of bipolar patients. Criteria for discontinuation during this study will be one or more of the following: 1) Missing more than five sessions during the Functional Remediation intervention 2) Hospitalization for any type of episode or clinical meaningful affective relapse 3) Withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I and II patients aged between 18 and 60.
* Three months of clinical remission.
* Patients will be required to present a moderate to severe degree of functional impairment (FAST>18).

Exclusion Criteria:

* IQ<85.
* Any medical condition that could affect neuropsychological performance.
* The presence of any comorbid psychiatric condition.
* Patients who received electroconvulsive therapy in the previous year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Psychosocial functioning measured by Functioning Assessment Short Test | 15 days
  The scale is interviewer-administered, designed for the assessment of psychosocial functioning. The 24 items of the scale are divided among 6 specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time. Each individual item is scored from 0 to 3. The global score (0-72) is obtained when the scores of each item are added up. The higher the score, the more serious the difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Torrent Font, PhD, Principal Investigator — Affiliated Postdoctoral Investigator
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sole B, Bonnin CM, Mayoral M, Amann BL, Torres I, Gonzalez-Pinto A, Jimenez E, Crespo JM, Colom F, Tabares-Seisdedos R, Reinares M, Ayuso-Mateos JL, Soria S, Garcia-Portilla MP, Ibanez A, Vieta E, Martinez-Aran A, Torrent C; CIBERSAM Functional Remediation Group. Functional remediation for patients with bipolar II disorder: improvement of functioning and subsyndromal symptoms. Eur Neuropsychopharmacol. 2015 Feb;25(2):257-64. doi: 10.1016/j.euroneuro.2014.05.010. Epub 2014 May 20. PMID 24906790
- [Background] Torrent C, Bonnin Cdel M, Martinez-Aran A, Valle J, Amann BL, Gonzalez-Pinto A, Crespo JM, Ibanez A, Garcia-Portilla MP, Tabares-Seisdedos R, Arango C, Colom F, Sole B, Pacchiarotti I, Rosa AR, Ayuso-Mateos JL, Anaya C, Fernandez P, Landin-Romero R, Alonso-Lana S, Ortiz-Gil J, Segura B, Barbeito S, Vega P, Fernandez M, Ugarte A, Subira M, Cerrillo E, Custal N, Menchon JM, Saiz-Ruiz J, Rodao JM, Isella S, Alegria A, Al-Halabi S, Bobes J, Galvan G, Saiz PA, Balanza-Martinez V, Selva G, Fuentes-Dura I, Correa P, Mayoral M, Chiclana G, Merchan-Naranjo J, Rapado-Castro M, Salamero M, Vieta E. Efficacy of functional remediation in bipolar disorder: a multicenter randomized controlled study. Am J Psychiatry. 2013 Aug;170(8):852-9. doi: 10.1176/appi.ajp.2012.12070971. PMID 23511717
- [Background] Martinez-Aran A, Torrent C, Sole B, Bonnin CM, Rosa AR, Sanchez-Moreno J, Vieta E. Functional remediation for bipolar disorder. Clin Pract Epidemiol Ment Health. 2011;7:112-6. doi: 10.2174/1745017901107010112. Epub 2011 Jun 6. PMID 21687565
- [Result] Bonnin CM, Torrent C, Vieta E, Martinez-Aran A. Restoring functioning in bipolar disorder: functional remediation. Harv Rev Psychiatry. 2014 Nov-Dec;22(6):326-30. doi: 10.1097/HRP.0000000000000062. PMID 25377603